CLINICAL TRIAL: NCT02657291
Title: Costoclavicular vs Paracoracoid Approach to Infraclavicular Brachial Plexus Block: a Feasibility Study
Acronym: CPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Dr., London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LawsonHRI
Record Dates: First submitted 2015-12-10; First posted 2016-01-15 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Upper Limb Injury
MeSH Terms: conditions — Arm Injuries | interventions — Ropivacaine; Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Costoclavicular (Experimental): Ultrasound-guided infraclavicular block using Ropivacaine 0.5% 35 mL using the costoclavicular approach
  Interventions: Drug: Ropivacaine; Device: Ultrasound
- Paracoracoid (Active Comparator): Ultrasound-guided infraclavicular block using Ropivacaine 0.5% 35 mL using the paracoracoid or standard approach
  Interventions: Drug: Ropivacaine; Device: Ultrasound

INTERVENTIONS:
Drug: Ropivacaine — Local anesthetic
  Other Names: Naropin
Device: Ultrasound — Ultrasound guided block

SUMMARY:
Patients for upper limb surgeries who are candidates for infraclavicular block will be screened. Two techniques of infraclavicular block will be compared. Measured outcomes are performance times, block onset times, patient satisfaction, quality of block, and requirement for supplementary analgesia.

DETAILED DESCRIPTION:
Infraclavicular brachial plexus block under ultrasound guidance is used for surgeries on the upper limb. Traditionally, the block is performed at the lateral infraclavicular fossa where the cords are variable in position relative to the axillary artery. A recently introduced technique is the costoclavicular approach where the cords are viewed as relatively more superficial and clustered together compared to the traditional technique. Those meeting the inclusion criteria and will consent to participate in the study will be randomized to have either an infraclavicular block in the paracoracoid approach (Group 1) or an infraclavicular block in the costoclavicular approach (Group 2). All groups will have the same injectable volume (35 mls) and local anesthetic concentration (ropivacaine 0.5%). There will be 35 study patients for each group for a total of 70 patients.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory elective surgery of the upper limb
* ASA (American Society of Anesthesiologists physical status classification system) 1-4
* Suitable for procedure to be carried out under infraclavicular block

Exclusion Criteria:

* Inability to give informed consent, Allergy to local anesthetics, morphine or fentanyl
* Ongoing major medical or psychiatric problems
* Narcotic abuse
* Peripheral neuropathy or major neurological problems
* Scarring in area of blockade
* Inability to co-operate with post-operative evaluation
* Major coagulopathy
* Pregnancy and breast-feeding
* Women of childbearing age who are not taking adequate contraceptive precautions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Block onset time | 1 hour
  From the time needle is removed from the patient's skin up to the time when block is considered adequate for surgery

SECONDARY OUTCOMES:
Procedure duration | 1 hour
  From the time the US probe touches the skin to the time the needle is removed
Quality of block | 1 hour
Patient satisfaction | 1 day
  Satisfaction score (VAS ranging from 0 = completely dissatisfied to 10 = completely satisfied)
Requirement for supplemental analgesia or anesthesia | 1 day
  Quality of block will be assessed if adequate for surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, Principal Investigator — Western University
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karmakar MK, Sala-Blanch X, Songthamwat B, Tsui BC. Benefits of the costoclavicular space for ultrasound-guided infraclavicular brachial plexus block: description of a costoclavicular approach. Reg Anesth Pain Med. 2015 May-Jun;40(3):287-8. doi: 10.1097/AAP.0000000000000232. No abstract available. PMID 25899958
- [Background] Bigeleisen P, Wilson M. A comparison of two techniques for ultrasound guided infraclavicular block. Br J Anaesth. 2006 Apr;96(4):502-7. doi: 10.1093/bja/ael024. Epub 2006 Feb 24. PMID 16500953
- [Background] Mosaffa F, Gharaei B, Rafeeyan M, Gachkar L. Comparing vertical and coracoid approaches for infraclavicular block in orthopedic surgery of the forearm and hand. J Clin Anesth. 2012 May;24(3):196-200. doi: 10.1016/j.jclinane.2011.07.013. Epub 2012 Apr 5. PMID 22484026
- [Background] Acar S, Gurkan Y, Solak M, Toker K. Coracoid versus lateral sagittal infraclavicular block. Acta Orthop Traumatol Turc. 2013;47(1):32-7. doi: 10.3944/aott.2013.2615. PMID 23549315